CLINICAL TRIAL: NCT05091216
Title: A Clinical Study on the Effects of Traditional Chinese Medicine Mouthwash Solutions on the Oral Health of Leprosy Patients in Taiwan
Brief Title: The Effects of Traditional Chinese Medicine Mouthwash Solutions on the Oral Health of Leprosy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo-Sheng Sanatorium (Other Government)
Responsible Party: Principal Investigator, Hsu Wei Hung, Director of chinese medicine, Lo-Sheng Sanatorium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TH-IRB-0021-0012
Record Dates: First submitted 2021-09-29; First posted 2021-10-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Leprosy; Hansen's Disease; Xerostomia; Plaque
Keywords: Leprosy; Hansen's disease (HD); traditional Chinese medicine mouthwash; oral health; xerostomia; Plaque Index, PLI
MeSH Terms: conditions — Leprosy; Xerostomia; Plaque, Amyloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine Mouthwash Group (Experimental): The subjects use traditional Chinese medicine mouthwash after three meals a day and before going to bed, four times a day for 7 consecutive days. After 7 days, record the PLI value and conduct a xerostomia questionnaire, and then retrieve the mouthwash bottle the remaining dose was checked to determine compliance. Those with significantly poor compliance were excluded from the experiment, and then the daily cleaning measures were resumed. The subjects still followed the way of mouthwash four times a day until the end of the 21st day after the xerostomia questionnaire.
  Interventions: Other: Traditional Chinese Medicine mouthwash
- Dilute 50 times of Traditional Chinese Medicine Mouthwash Group (Active Comparator): The subjects use dilute 50 times traditional Chinese medicine mouthwash after three meals a day and before going to bed, four times a day for 7 consecutive days. After 7 days, record the PLI value and conduct a xerostomia questionnaire, and then retrieve the mouthwash bottle the remaining dose was checked to determine compliance. Those with significantly poor compliance were excluded from the experiment, and then the daily cleaning measures were resumed. The subjects still followed the way of mouthwash four times a day until the end of the 21st day after the xerostomia questionnaire.
  Interventions: Other: Dilute 50 times of Traditional Chinese Medicine mouthwash

INTERVENTIONS:
Other: Traditional Chinese Medicine mouthwash — The mouthwash used in this test is based on the records of past traditional Chinese medicine classics and the existing antibacterial experimental evidence. The selected medicinal materials are honeysuckle, scutellaria, peppermint, licorice, and rhizome.
  Arms: Traditional Chinese Medicine Mouthwash Group
Other: Dilute 50 times of Traditional Chinese Medicine mouthwash — Dilute 50 times of traditional Chinese medicine mouthwash.
  Arms: Dilute 50 times of Traditional Chinese Medicine Mouthwash Group

SUMMARY:
The purpose of this study is to treat with traditional Chinese medicine mouthwash, and through the research of dental plaque detection and xerostomia questionnaire and traditional Chinese medicine treatment mechanism.

DETAILED DESCRIPTION:
The study will recruit 58 patients who are hospitalized at Lo-Sheng Sanatorium, Ministry of Health and Welfare. Investigators will use xerostomia questionnaire and PLI examination to collect the subject's data. Separate subjects in to two group randomly. The control group will use the traditional Chinese medicine mouthwash, and the other group will use the dilute 50 times of traditional Chinese medicine mouthwash.

Every 7 days will record the PLI value and conduct a xerostomia questionnaire, until 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Lo-Sheng sanatorium of the Ministry of Health and Welfare, Taiwan
* Compliant with the presence of more than four teeth in each of the upper and lower four regions
* Those who have not used antibiotics and mouthwash two months before the test

Exclusion Criteria:

* Moderate to severe dementia
* CDR (Clinical Dementia Assessment Scale) is greater than or equal to 2 points or more
* Those with a score of less than 17 on the MMSE Simple Mind Scale
* Nasogastric Tube Inserters
* Those who are allergic to mouthwash
* Those who are on course of antibiotics and steroids
* Those who have had dental cleansing within one month

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Plaque Index, PLI | 21 days
  Turesky modification of the Quigley-Hein Plaque Index (TQHPI)
Xerostomia questionnaire | 21 days
  Xerostomia questionnaire, Pai (2001)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Hung Hsu, Principal Investigator — Lo-Sheng Sanatorium
Locations (1):
- Lo-Sheng Sanatorium, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-09-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT05091216/Prot_ICF_000.pdf